CLINICAL TRIAL: NCT00944957
Title: Patient Preference, Sleep Quality, and Anxiety/Depression: Comparison of Raltegravir and Efavirenz
Brief Title: Patient Preference, Sleep Quality, and Anxiety/Depression: A Comparison of Raltegravir and Efavirenz
Acronym: Switch-ER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Bern (Other); University of Lausanne Hospitals (Other); Hospital Lugano (Unknown); University Hospital, Basel, Switzerland (Other); Hospital of Neuchâtel (Unknown); University Hospital, Zürich (Other)
Responsible Party: Professeur Bernard Hirschel, Geneva infectious diseases
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IEC 09-087
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-07

CONDITIONS: Sleep Disorders; HIV Infections
Keywords: Raltegravir; efavirenz; anxiety; depression; sleep quality; HIV; NNRTI; Tritherapy; compliance; stocrin; treatment experienced
MeSH Terms: conditions — Sleep Wake Disorders; HIV Infections; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Patient Compliance | interventions — Raltegravir Potassium; efavirenz

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir first (Experimental): Patients treated with Raltegravir for first 2 weeks
  Interventions: Drug: Raltegravir for the first 2 weeks; Drug: Efavirenz for the last 2 weeks
- Efavirenz first (Experimental): Patients treated with Efavirenz for first 2 weeks
  Interventions: Drug: Efavirenz for the first 2 weeks; Drug: Raltegravir for the last 2 weeks

INTERVENTIONS:
Drug: Raltegravir for the first 2 weeks — Patient receives raltegravir and efavirenz placebo during the first 2 weeks
  Arms: Raltegravir first
Drug: Efavirenz for the last 2 weeks — Patient receives efavirenz and raltegravir placebo during the last 2 weeks
  Arms: Raltegravir first
Drug: Efavirenz for the first 2 weeks — Efavirenz and raltegravir placebo for the first 2 weeks
  Arms: Efavirenz first
Drug: Raltegravir for the last 2 weeks — Raltegravir and efavirenz placebo for the last 2 weeks
  Arms: Efavirenz first

SUMMARY:
Efavirenz causes neuropsychiatric side effects and sleep disturbance, including vivid dreams, dizziness, and abnormal tiredness. These symptoms are frequent during the first weeks of treatment, with subsequent attenuation but may not completely resolve even years after efavirenz initiation.

The investigators plan a four week, randomized, placebo-controlled, double-blind study. In group 1, efavirenz will be replaced with efavirenz placebo plus raltegravir, in group 2, efavirenz would be continued, and raltegravir placebo given in addition. After two weeks, patients in group 1 would switch to the regimen of group 2, and vice versa.

The primary endpoint of the trial will be patient preference. Sleep quality, daytime sleepiness, and anxiety will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years
* Signing the study consent form and agree to change ART regimen
* Stable HAART including EFV since at least 3 months
* HIV-RNA below 50 copies for at least 3 months

Exclusion Criteria:

* No major psychiatric disease (psychosis, severe depression) diagnosed before the initiation of EFV
* Mentally incompetent patients
* Pregnancy or lactation Women of childbearing potential must use one or two reliable contraceptive methods during the trial, from day 1 to the end of week 12. Acceptable methods include the birth control pill, IUD, condoms with spermicides. Non-acceptable methods include (non-exhaustive list): Withdrawal, calendar (Onigo method), or spermicides alone.
* Concomitant renal or hepatic disease:

  * Creatinine above 150 micromol/L
  * Transaminases above 5 times upper normal limit
  * Prothrombin (Quick) value below 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2009-12 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Symptoms and neurological side effects of study drugs | baseline, week 2 and week 4

SECONDARY OUTCOMES:
Levels of daytime sleepiness | baseline, week 2 and week 4
Sleep Quality | baseline, week 2 and week 4
Patient preference | 4 weeks
Symptoms of depression, anxiety and stress will be assessed | baseline, week 2 and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Bernard BH Hirschel, Professor, Principal Investigator — Geneva Hospital
Locations (1):
- University Hopistal of Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- See also: Swiss HIV Cohort Study — http://www.shcs.ch